CLINICAL TRIAL: NCT00942357
Title: A Randomized Phase III Trial of Cisplatin and Tumor Volume Directed Irradiation Followed by Carboplatin and Paclitaxel vs. Carboplatin and Paclitaxel for Optimally Debulked, Advanced Endometrial Carcinoma
Brief Title: Carboplatin and Paclitaxel With or Without Cisplatin and Radiation Therapy in Treating Patients With Stage I, Stage II, Stage III, or Stage IVA Endometrial Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0258; NCI-2011-01951 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-00685; CDR0000649079; GOG-0258 (Other: NRG Oncology); GOG-0258 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Stage IA Uterine Corpus Cancer AJCC v7; Stage IB Uterine Corpus Cancer AJCC v7; Stage II Uterine Corpus Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Brachytherapy; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cisplatin, radiation therapy, paclitaxel, carboplatin) (Experimental): Patients receive cisplatin IV on days 1 and 29. Patients also undergo radiation therapy QD, 5 days a week, for 5-6 weeks. Some patients may then undergo brachytherapy over 2-3 weeks. Beginning within 8 weeks after completion of chemoradiotherapy, patients receive paclitaxel IV over 3 hours and carboplatin IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Radiation: Internal Radiation Therapy; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy
- Arm II (paclitaxel and carboplatin) (Active Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (cisplatin, radiation therapy, paclitaxel, carboplatin)
Radiation: Internal Radiation Therapy — Undergo brachytherapy
  Other Names: BRACHYTHERAPY; internal radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
  Arms: Arm I (cisplatin, radiation therapy, paclitaxel, carboplatin)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Arm I (cisplatin, radiation therapy, paclitaxel, carboplatin)

SUMMARY:
This randomized phase III trial studies carboplatin and paclitaxel to see how well they work with or without cisplatin and radiation therapy in treating patients with stage I-IVA endometrial cancer. Drugs used in chemotherapy, such as carboplatin, paclitaxel, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether carboplatin and paclitaxel are more effective with or without cisplatin and radiation therapy in treating patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if treatment with cisplatin and volume-directed radiation followed by carboplatin and paclitaxel for 4 cycles (experimental arm) reduces the rate of recurrence or death (i.e., increases recurrence-free survival) when compared to chemotherapy consisting of carboplatin and paclitaxel for 6 cycles (control arm) in patients with stages III-IVA endometrial carcinoma (< 2 cm residual disease) or patients with International Federation of Gynecology and Obstetrics (FIGO) 2009 stage I or II serous (uterine papillary serous carcinoma [UPSC]) or clear cell endometrial carcinoma and positive cytology.

SECONDARY OBJECTIVES:

I. To determine if treatment with cisplatin and volume-directed radiation followed by carboplatin and paclitaxel for 4 cycles (experimental arm) reduces the rate of death (i.e., increases survival) when compared to chemotherapy consisting of carboplatin and paclitaxel for 6 cycles (control arm) in patients with stages III-IVA endometrial carcinoma (< 2 cm residual disease) or patients with FIGO 2009 stage I or II serous (UPSC) or clear cell endometrial carcinoma and positive cytology.

II. To compare the regimens with respect to acute and late adverse effects of therapy.

III. To determine the impact of patient-reported quality of life during and following treatment for up to 1 year with the two treatment regimens.

TERTIARY OBJECTIVES:

I. To bank formalin-fixed, paraffin-embedded (FFPE) tumor tissue and whole blood specimens for future research.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cisplatin intravenously (IV) on days 1 and 29. Patients also undergo radiation therapy once daily (QD), 5 days a week, for 5-6 weeks. Some patients may then undergo brachytherapy over 2-3 weeks. Beginning within 8 weeks after completion of chemoradiotherapy, patients receive paclitaxel IV over 3 hours and carboplatin IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel IV over 3 hours and carboplatin IV on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients with surgical stage III or IVA endometrial carcinoma per FIGO 2009 staging criteria including clear cell and serous papillary and undifferentiated carcinoma

  * Surgical stage III disease includes those patients with positive adnexa, parametrial involvement, tumor invading the serosa, positive pelvic and/or para-aortic nodes, or vaginal involvement
  * Surgical stage IVA patients with bladder or bowel mucosal involvement, but no spread outside the pelvis
* Patients with FIGO 2009 surgical stage I or II endometrial clear cell or serous carcinoma and with positive peritoneal cytology
* Surgery must have included a hysterectomy and bilateral salpingo-oophorectomy; pelvic lymph node sampling and para-aortic lymph node sampling are optional
* Patients with a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* White blood cell (WBC) >= 3,000/mcl
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 2.5 x upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 times ULN
* Bilirubin =< 1.5 times ULN
* Creatinine =< institutional ULN
* Patients who have met the pre-entry requirements; testing values/results must meet eligibility criteria
* Patients who have signed an approved informed consent and authorization permitting release of personal health information
* Entry into the study is limited to no more than 8 weeks from the date of surgery

Exclusion Criteria:

* Patients with carcinosarcoma
* Patients with recurrent endometrial cancer
* Patients with residual tumor after surgery (any single site) exceeding 2 cm in maximum dimension
* Patients who have had pelvic or abdominal radiation therapy
* Patients with positive pelvic washings as the only extra-uterine disease are NOT eligible if the histology is other than clear cell or papillary serous carcinoma
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of active malignancy within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients with a history of serious co-morbid illness or uncontrolled illnesses that would preclude protocol therapy
* Patients with an estimated survival of less than three months
* Patients with FIGO 2009 stage IVB endometrial cancer
* Patients with parenchymal liver metastases
* Patients who have received prior chemotherapy for endometrial cancer
* Patients with a history of myocardial infarction, unstable angina, or uncontrolled arrhythmia within 3 months from enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2009-06-29 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2024-07-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela E Matei, Principal Investigator — NRG Oncology
Locations (670):
- United States (655):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Tennessee Valley Gynecologic Oncology, Huntsville, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Gynecologic Oncology Associates-Newport Beach, Newport Beach, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Southeast Gynecologic Oncology Associates, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Mercy Hospital, Miami, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Saint Margaret Health-Dyer Campus, Dyer, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Saint Margaret Health-Hammond Campus, Hammond, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Abben Cancer Center, Spencer, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Willis-Knighton Medical and Cancer Center, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Tennessee Oncology PLLC- Centennial Medical Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (5):
  - McGill University Department of Oncology, Montreal, Quebec
  - McGill University Health Centre at Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Saint Mary's Hospital, Montreal, Quebec
- South Korea (10):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Korea
  - Catholic University of Korea-Seoul Saint Mary's Hospital, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Matei DE, Enserro DM, Randall ME, Mutch D, Small W, DiSilvestro PA, Spirtos NM, O'Malley DM, Cantuaria GH, Michelin D, Waggoner S, Shahin M, Guntupalli S, Lara O, Ueland FR, Warshal D, Bonebrake A, Tewari KS, Tan A, Powell MA, Walker JL, Santin AD, Kim JH, Miller DS. Long-Term Follow-Up and Overall Survival in NRG258, a Randomized Phase III Trial of Chemoradiation Versus Chemotherapy for Locally Advanced Endometrial Carcinoma. J Clin Oncol. 2025 Mar 20;43(9):1055-1060. doi: 10.1200/JCO.24.01121. Epub 2024 Dec 19. PMID 39700442
- [Derived] Matulonis UA, Huang HQ, Filiaci VL, Randall M, DiSilvestro PA, Moxley KM, Fowler JM, Powell MA, Spirtos NM, Tewari KS, Richards WE, Nakayama JM, Mutch DG, Miller DS, Matei D, Wenzel LB. Patient reported outcomes for cisplatin and radiation followed by carboplatin/paclitaxel versus carboplatin/paclitaxel for locally advanced endometrial carcinoma: An NRG oncology study. Gynecol Oncol. 2022 Feb;164(2):428-436. doi: 10.1016/j.ygyno.2021.11.021. Epub 2021 Dec 11. PMID 34903380
- [Derived] Matei D, Filiaci V, Randall ME, Mutch D, Steinhoff MM, DiSilvestro PA, Moxley KM, Kim YM, Powell MA, O'Malley DM, Spirtos NM, Small W Jr, Tewari KS, Richards WE, Nakayama J, Matulonis UA, Huang HQ, Miller DS. Adjuvant Chemotherapy plus Radiation for Locally Advanced Endometrial Cancer. N Engl J Med. 2019 Jun 13;380(24):2317-2326. doi: 10.1056/NEJMoa1813181. PMID 31189035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 0258 accrued 813 patients between June 29, 2009 and July 28, 2014.
Period: Overall Study
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
Started | 407 | 406
Completed | 370 | 366
Not Completed | 37 | 40
Not completed — Ineligible | 37 | 40

BASELINE CHARACTERISTICS:
Population: All eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin) | Total
Number analyzed (Participants) | 370 | 366 | 736
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 0 | 0
  30-39 years | 6 | 10 | 16
  40-49 years | 36 | 31 | 67
  50-59 years | 132 | 136 | 268
  60-69 years | 133 | 130 | 263
  70-79 years | 55 | 51 | 106
  80-89 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370 | 366 | 736
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 29 | 44
  Not Hispanic or Latino | 338 | 324 | 662
  Unknown or Not Reported | 17 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 33 | 34 | 67
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 37 | 42 | 79
  White | 291 | 279 | 570
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Endometrial Cancer Grades [Count of Participants; unit: Participants] — Grade 1 is 5% or less of a non-squamous or non-morular solid growth pattern. Grade 2 is 6 through 50% of a non squamous or non-morular solid growth pattern. Grade 3 is more than 50% of a non-squamous or non-morular solid growth pattern. Generally the higher the stage the worse the outcome.
  Participants
    Endometrioid Grade 1 | 87 | 79 | 166
    Endometrioid Grade 2 | 103 | 118 | 221
    Endometrioid Grade 3 | 66 | 62 | 128
    Serous | 66 | 65 | 131
    Clear Cell | 10 | 12 | 22
    Other | 38 | 30 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence, Progression or Death
Description: Number of participants enrolled with recurrence or progression of disease or death up to date of last contact. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions.
Time Frame: Disease was to be assessed at baseline, end of treatment and every 6 months for two years, and annually up to 5 years.
Population: Number of recurrence, progression or death events in eligible and enrolled patients
Measure: Number; unit: participants
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
Number analyzed (Participants) | 370 | 366
participants | 132 | 139

2. Secondary Outcome: Number of Participants With Acute Adverse Effects as Graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version (CTCAE) Version 3.0
Description: The maximum grade of all treatment emergent adverse events without regard to attribution. General guidelines for severity of adverse events are as follows: Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life threatening and Grade 5 is death.
Time Frame: Assessed throughout the treatment period and for 21-30 days after discontinuation of treatment
Population: Eligible and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
Number analyzed (Participants) | 346 | 361
Participants
  Grade 1 | 5 | 15
  Grade 2 | 139 | 118
  Grade 3 | 154 | 119
  Grade 4 | 48 | 105
  Grade 5 | 0 | 3

3. Secondary Outcome: Number of Participants With Late Adverse Events as Graded by the NCI CTCAE Version 3.0
Description: The maximum grade of Adverse events reported during follow-up until progression of disease, a change of therapy or otherwise off study for a maximum of 3 years without regard to attribution. General guidelines for severity of adverse events are as follows: Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life threatening and Grade 5 is death.
Time Frame: Assessed every 6 months for 3 years
Population: All eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
Number analyzed (Participants) | 346 | 361
Participants
  Grade 1 | 85 | 96
  Grade 2 | 71 | 79
  Grade 3 | 45 | 33
  Grade 4 | 14 | 7
  Grade 5 | 1 | 4

4. Secondary Outcome: Overall Survival
Description: Independence between the two endpoints, RFS and survival, and randomized treatment will be assessed with a stratified logrank test for an intent-to-treat analysis of eligible patients.
Time Frame: From entry into the study to death or the date of last contact, assessed up to 8 years
Reporting Status: Not Posted

5. Secondary Outcome: Patient-reported Peripheral Neuropathy Symptoms
Description: Patient reported peripheral neuropathy symptoms was measured with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The FACT/GOG-Ntx subscale contains 4 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative items, reversal was performed prior to score calculation. According to the FACIT measurement system, the Ntx score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The Ntx score ranges 0-16 with a large score suggests less peripheral neuropathy symptoms.
Time Frame: Prior to study treatment (baseline), Arm 1: 1 week post completion of radiation therapy, Arm 2: Prior to cycle 3 (6 weeks post starting of study treatment), 18 weeks post the starting of study treatement, 70 weeks post the starting of study treatment
Population: Patients who provided baseline and >= 1 follow-up assessment(s)
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
Number analyzed (Participants) | 332 | 349
unit on a scale
  Baseline | 14.9 (0.1) | 15.0 (0.1)
  6 weeks | 14.4 (0.4) | 12.4 (0.4)
  18 weeks | 10.4 (0.4) | 9.9 (0.5)
  70 weeks | 11.8 (0.4) | 11.6 (0.4)

6. Secondary Outcome: Patient-reported Quality of Life (QOL)
Description: Patient reported quality of life was measured with the Treatment Outcome Index of the Functional Assessment of Cancer Therapy for endometrial cancer (FACT-En TOI). It is a scale for assessing general QOL of endometrial cancer patients. It consists of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Endometrium Cancer subscale (16 items). Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). According to the FACIT measurement system, a subscale score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the subscale. The FACT-En TOI score is calculated as the sum of the subscale scores, ranges are 0-120 with a large score suggesting a better QOL.
Time Frame: Prior to study treatment (baseline), Arm 1: 1 Week post completion of radiation therapy, Arm 2: Prior to cycle 3 (6 weeks post starting of study treatment), 18 weeks post the starting of study treatment, 70 weeks post the starting of study treatment
Population: Patients who provided baseline and >= 1 follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
Number analyzed (Participants) | 332 | 349
units on a scale
  Baseline | 98.4 (0.8) | 97.6 (0.8)
  6 weeks | 89.5 (2.1) | 90.9 (2.0)
  18 weeks | 87.8 (2.1) | 93.0 (2.0)
  70 weeks | 96.0 (2.2) | 99.4 (2.1)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Description: All-Cause Mortality will be reported at the end of the study after final data collection is complete. The number currently listed (0) is indicating the data collection is incomplete. The number reported differs from the participant flow because some of the participants were not treated. The number reported are eligible and treated.
Arm/Group | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) | Arm II (Paclitaxel and Carboplatin)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 78/346 | 61/361
Other Adverse Events (participants affected / at risk) | 346/346 | 360/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) (N=346) | Arm II (Paclitaxel and Carboplatin) (N=361)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 3 | 2
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 | 1
Neutrophils (Blood and lymphatic system disorders) | 5 | 27
Platelets (Blood and lymphatic system disorders) | 0 | 2
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 6 | 0
Hemoglobin (Blood and lymphatic system disorders) | 4 | 2
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 2 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 0 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 1 | 1
Fever (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Death No Ctcae Term - Disease Progression Nos (General disorders) | 0 | 1
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Rectum (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 9 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1 | 0
Febrile Neutropenia (Infections and infestations) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Blood (Infections and infestations) | 1 | 2
Infection - Other (Infections and infestations) | 3 | 1
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Lymphatic (Infections and infestations) | 0 | 1
Inf Unknown Anc: Kidney (Infections and infestations) | 0 | 1
Inf Unknown Anc: Wound (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Pelvis Nos (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 1 | 0
Alt (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Psychosis (Nervous system disorders) | 1 | 0
Neurology - Other (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Pain: Head/Headache (General disorders) | 1 | 0
Pain: Back (General disorders) | 2 | 0
Pain: Abdominal Pain Nos (General disorders) | 1 | 2
Pain: Cardiac/ Heart (General disorders) | 1 | 1
Pain: Neuralgia (General disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 3 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cisplatin, Radiation Therapy, Paclitaxel, Carboplatin) (N=346) | Arm II (Paclitaxel and Carboplatin) (N=361)
Allergy/Immunology - Other (Immune system disorders) | 3 | 2
Allergic Reaction/Hypersensitivity (Immune system disorders) | 15 | 28
Rhinitis (Immune system disorders) | 7 | 15
Autoimmune Reaction (Immune system disorders) | 0 | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 2 | 2
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 4 | 2
Tinnitus (Ear and labyrinth disorders) | 18 | 13
Neutrophils (Blood and lymphatic system disorders) | 176 | 246
Platelets (Blood and lymphatic system disorders) | 217 | 195
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 12 | 19
Bone Marrow Cellularity (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 287 | 262
Lymphopenia (Blood and lymphatic system disorders) | 53 | 21
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 309 | 292
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 14 | 7
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 3 | 0
S/N Arrhythmia: Atrial Flutter (Cardiac disorders) | 1 | 0
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 11 | 8
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1 | 0
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 0 | 1
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 24 | 46
Valvular Heart Disease (Cardiac disorders) | 1 | 0
Cardiac General - Other (Cardiac disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Hypotension (Cardiac disorders) | 6 | 10
Inr (Vascular disorders) | 1 | 6
Coagulopathy - Other (Vascular disorders) | 0 | 1
Ptt (Vascular disorders) | 0 | 3
Constitutional Symptoms - Other (General disorders) | 11 | 13
Sweating (General disorders) | 10 | 8
Weight Gain (General disorders) | 6 | 15
Fever (General disorders) | 28 | 14
Weight Loss (General disorders) | 41 | 12
Obesity (General disorders) | 1 | 0
Rigors/Chills (General disorders) | 16 | 15
Fatigue (General disorders) | 294 | 271
Insomnia (General disorders) | 56 | 63
Nail Changes (Skin and subcutaneous tissue disorders) | 9 | 14
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 208 | 258
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 2 | 3
Dermatitis - Chemoradiation (Skin and subcutaneous tissue disorders) | 3 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Cheilitis (Skin and subcutaneous tissue disorders) | 0 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1 | 2
Bruising (Skin and subcutaneous tissue disorders) | 8 | 5
Acne (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 48 | 44
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 13
Dermatitis - Radiation (Skin and subcutaneous tissue disorders) | 17 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 19
Burn (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 4
Flushing (Skin and subcutaneous tissue disorders) | 11 | 10
Hand-Foot (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 18 | 14
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 5
Ulceration (Skin and subcutaneous tissue disorders) | 5 | 1
Hot Flashes (Endocrine disorders) | 38 | 38
Diabetes (Endocrine disorders) | 1 | 0
Endocrine - Other (Endocrine disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 6 | 0
Flatulence (Gastrointestinal disorders) | 8 | 5
Ulcer,gi - Stoma (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 13 | 3
Heartburn (Gastrointestinal disorders) | 27 | 22
Dental: Teeth (Gastrointestinal disorders) | 0 | 1
Mucositis (Functional/Sympt) - Pharynx (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Leak, Gi - Rectum (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 7
Distention (Gastrointestinal disorders) | 15 | 7
Taste Alteration (Gastrointestinal disorders) | 34 | 38
Incontinence, Anal (Gastrointestinal disorders) | 3 | 1
Fistula, Gi - Abdomen Nos (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 10 | 9
Mucositis (Functional/Sympt) - Rectum (Gastrointestinal disorders) | 2 | 0
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 14 | 17
Colitis (Gastrointestinal disorders) | 0 | 2
Mucositis (Clinical Exam) - Rectum (Gastrointestinal disorders) | 1 | 0
Mucositis (Functional/Sympt) - Anus (Gastrointestinal disorders) | 1 | 0
Dentures (Gastrointestinal disorders) | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 14 | 18
Vomiting (Gastrointestinal disorders) | 104 | 76
Anorexia (Gastrointestinal disorders) | 121 | 84
Dehydration (Gastrointestinal disorders) | 29 | 11
Constipation (Gastrointestinal disorders) | 139 | 173
Nausea (Gastrointestinal disorders) | 235 | 183
Gastrointestinal - Other (Gastrointestinal disorders) | 13 | 5
Diarrhea (Gastrointestinal disorders) | 253 | 95
Mucositis (Clinical Exam) - Pharynx (Gastrointestinal disorders) | 0 | 1
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 5 | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 6 | 6
Hemorrhage, Gi - Rectum (Vascular disorders) | 7 | 6
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 6 | 5
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 1 | 0
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 1 | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 1 | 1
Hemorrhage, Gi - Colon (Vascular disorders) | 0 | 1
Hemorrhage, Cns (Vascular disorders) | 1 | 0
Petechiae (Vascular disorders) | 1 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 | 1
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Wound (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 3
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Neck Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 6 | 5
Febrile Neutropenia (Infections and infestations) | 3 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Rectum (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 19 | 14
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 1 | 0
Inf Unknown Anc: Blood (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 16 | 9
Opportunisitic Inf Assoc. W/Gr 2 Lymphopenia (Infections and infestations) | 2 | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 2 | 0
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 0 | 1
Inf Unknown Anc: Vulva (Infections and infestations) | 1 | 1
Inf Unknown Anc: Vagina (Infections and infestations) | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Mucosa (Infections and infestations) | 1 | 0
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 3 | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 1 | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Bronchus (Infections and infestations) | 1 | 0
Inf Unknown Anc: Soft Tissue Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc:peritoneal Cavity (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 13 | 12
Inf Unknown Anc: Urethra (Infections and infestations) | 0 | 1
Inf Unknown Anc: Kidney (Infections and infestations) | 1 | 0
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1 | 1
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 1
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Joint (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Lymphatic (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 3 | 3
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 4
Inf W/Gr 3 Or 4 Anc: Urethra (Infections and infestations) | 0 | 1
Lymphatics - Other (Blood and lymphatic system disorders) | 0 | 1
Lymphocele (Blood and lymphatic system disorders) | 1 | 2
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 2 | 1
Edema: Limb (Blood and lymphatic system disorders) | 56 | 51
Edema: Head And Neck (Blood and lymphatic system disorders) | 2 | 3
Ast (Metabolism and nutrition disorders) | 23 | 34
Gfr (Metabolism and nutrition disorders) | 4 | 4
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 8 | 9
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Cholesterol,serum High (Metabolism and nutrition disorders) | 0 | 2
Proteinuria (Metabolism and nutrition disorders) | 5 | 1
Hemoglobinuria (Metabolism and nutrition disorders) | 2 | 0
Creatinine (Metabolism and nutrition disorders) | 39 | 24
Hypoalbuminemia (Metabolism and nutrition disorders) | 29 | 33
Ggt (Metabolism and nutrition disorders) | 2 | 0
Alt (Metabolism and nutrition disorders) | 28 | 33
Alkaline Phosphatase (Metabolism and nutrition disorders) | 40 | 35
Bilirubin (Metabolism and nutrition disorders) | 5 | 5
Lipase (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatremia (Metabolism and nutrition disorders) | 39 | 31
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 3 | 0
Hypernatremia (Metabolism and nutrition disorders) | 7 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 35 | 20
Hyperkalemia (Metabolism and nutrition disorders) | 14 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 78 | 73
Hypokalemia (Metabolism and nutrition disorders) | 50 | 44
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 70 | 53
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 8 | 10
Lumbar Spine Rom (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint-Function (Musculoskeletal and connective tissue disorders) | 0 | 3
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Gait/Walking (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 8
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 36 | 19
Muscle Weakness - Right-Sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 18 | 11
Syncope (Nervous system disorders) | 2 | 3
Involuntary Movement (Nervous system disorders) | 3 | 3
Psychosis (Nervous system disorders) | 0 | 2
Neurology - Other (Nervous system disorders) | 8 | 9
Mental Status (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Mood Alteration - Euphoria (Nervous system disorders) | 0 | 2
Mood Alteration - Depression (Nervous system disorders) | 35 | 37
Mood Alteration - Anxiety (Nervous system disorders) | 35 | 41
Mood Alteration - Agitation (Nervous system disorders) | 1 | 7
Tremor (Nervous system disorders) | 5 | 5
Speech Impairment (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 2 | 1
Personality (Nervous system disorders) | 1 | 0
Irritability (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 3 | 6
Ataxia (Nervous system disorders) | 3 | 2
Confusion (Nervous system disorders) | 4 | 4
Memory Impairment (Nervous system disorders) | 10 | 12
Dizziness (Nervous system disorders) | 40 | 57
Neuropathy,cranial - Cn Viii Hearing/Balance (Nervous system disorders) | 1 | 0
Neuropathy,cranial - Cn I Smell (Nervous system disorders) | 1 | 0
Neuropathy-Sensory (Nervous system disorders) | 230 | 253
Neuropathy-Motor (Nervous system disorders) | 11 | 21
Retinopathy (Eye disorders) | 0 | 1
Ocular/Visual - Other (Eye disorders) | 3 | 2
Vitreous Hemorrhage (Eye disorders) | 1 | 0
Watery Eye (Eye disorders) | 1 | 3
Dry Eye (Eye disorders) | 3 | 1
Ocular Surface Disease (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Photophobia (Eye disorders) | 2 | 0
Flashing Lights/Floaters (Eye disorders) | 3 | 6
Diplopia (Eye disorders) | 0 | 2
Blurred Vision (Eye disorders) | 19 | 25
Pain - Other (General disorders) | 24 | 18
Pain: Urethra (General disorders) | 15 | 2
Pain: Perineum (General disorders) | 4 | 0
Pain: Pelvis (General disorders) | 8 | 11
Pain: Breast (General disorders) | 0 | 1
Pain: Vagina (General disorders) | 8 | 2
Pain: Chest /Thorax Nos (General disorders) | 10 | 7
Pain: Chest Wall (General disorders) | 3 | 2
Pain: Throat/Pharynx/Larynx (General disorders) | 5 | 6
Pain: Larynx (General disorders) | 1 | 1
Pain: Eye (General disorders) | 2 | 0
Pain: Head/Headache (General disorders) | 42 | 56
Pain: Neck (General disorders) | 2 | 1
Pain: Intestine (General disorders) | 2 | 0
Pain: Extremity-Limb (General disorders) | 48 | 63
Pain: Buttock (General disorders) | 3 | 1
Pain: Back (General disorders) | 25 | 34
Pain: Joint (General disorders) | 76 | 102
Pain: Bone (General disorders) | 68 | 40
Pain: Gallbladder (General disorders) | 1 | 0
Pain: Kidney (General disorders) | 1 | 0
Pain: Bladder (General disorders) | 16 | 3
Pain: Pain Nos (General disorders) | 9 | 8
Pain: Stomach (General disorders) | 2 | 2
Pain: Rectum (General disorders) | 5 | 0
Pain: Peritoneum (General disorders) | 1 | 0
Pain: Oral Cavity (General disorders) | 3 | 2
Pain: Esophagus (General disorders) | 2 | 0
Pain: Dental/Teeth/Peridontal (General disorders) | 3 | 2
Pain: Abdominal Pain Nos (General disorders) | 79 | 53
Pain: Scalp (General disorders) | 2 | 5
Pain: Oral - Gums (General disorders) | 0 | 4
Pain: Skin (General disorders) | 3 | 0
Pain: Middle Ear (General disorders) | 0 | 1
Pain: Cardiac/ Heart (General disorders) | 0 | 2
Pain: Muscle (General disorders) | 67 | 82
Pain: Anus (General disorders) | 3 | 0
Pain: Neuralgia (General disorders) | 2 | 2
Pain: Sinus (General disorders) | 1 | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Edema, Larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 45
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 76 | 65
Renal/Genitourinary - Other (Renal and urinary disorders) | 19 | 5
Leak, Gu - Vagina (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 19 | 4
Urinary Color Change (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 6 | 4
Obstruction, Gu - Ureter (Renal and urinary disorders) | 2 | 1
Obstruction, Gu - Stoma (Renal and urinary disorders) | 1 | 0
Obstruction, Gu - Bladder (Renal and urinary disorders) | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 35 | 14
Bladder Spasm (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 61 | 21
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast (Reproductive system and breast disorders) | 2 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 4 | 2
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 3 | 4
Vaginitis (Reproductive system and breast disorders) | 2 | 1
Vaginal Stenosis (Reproductive system and breast disorders) | 4 | 0
Vaginal Mucositis (Reproductive system and breast disorders) | 5 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 12 | 7
Orgasmic Function (Reproductive system and breast disorders) | 0 | 1
Intra-Op Injury: Urinary Tract Nos (Surgical and medical procedures) | 1 | 0
Intra-Op Injury: Other (Surgical and medical procedures) | 1 | 0
Syndromes - Other (General disorders) | 1 | 1
Cytokine Release Syndrome (General disorders) | 0 | 1
Flu-Like Syndrome (General disorders) | 1 | 8
Vascular - Other (Vascular disorders) | 2 | 0
Portal Flow (Vascular disorders) | 1 | 0
Artery Injury - Visceral (Vascular disorders) | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6 | 9
Phlebitis (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT00942357/Prot_SAP_000.pdf